CLINICAL TRIAL: NCT00295581
Title: Phase 1 Study of the Safety and Immunogenicity of PpPfs25/ISA51 and ScPvs25/ISA51: Transmission Blocking Vaccines for Plasmodium Falciparum and Plasmodium Vivax Malaria
Brief Title: PpPfs25/ISA51 and ScPvs25/ISA51 Vaccines for Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050118; 05-I-0118
Record Dates: First submitted 2006-02-23; First posted 2006-02-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-17

CONDITIONS: Plasmodium Falciparum; Plasmodium Vivax Malaria
Keywords: Human; Clinical Trial; Mosquito; Healthy Volunteer; HV
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax

INTERVENTIONS:
Drug: PpPfs25/ISA51 & ScPvs25/ISA51

SUMMARY:
This study, conducted at Johns Hopkins University Center for Immunization Research in Washington DC, will test the safety and immune response of healthy volunteers to two experimental malaria vaccines. Malaria is a disease of red blood cells caused by a parasite that spreads from person to person by mosquitoes. It affects people of all ages, but is particularly severe in children. Patients may have a high fever, chills and muscle aches. They sometimes can have severe complications that may even result in death.

The vaccines in this study are called "transmission blocking" vaccines. These vaccines stimulate the person's immune system to produce antibodies against malaria. When a mosquito bites a vaccinated person, it ingests some of the person's blood. The antibodies in the ingested blood stop the malaria parasite from developing inside the mosquito. The mosquito would not be able to transmit malaria to other people. PpPfs25/ISA51 (Vaccine A) stimulates production of antibodies against the malaria parasite Plasmodium falciparum, and ScPvs25/ISA51 (Vaccine B) stimulates antibodies against the malaria parasite Plasmodium vivax. The vaccines also contain a substance called Montanide ISA51, which boosts the immune response to the vaccine.

Healthy volunteers between 18 and 50 years of age may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests. Women who are able to become pregnant have a urine pregnancy test before each immunization.

Participants are randomly assigned to receive two injections, spaced 4 months apart, of either Vaccine A or Vaccine B at one of three doses-high, medium, or low. Two subjects in each dose group additionally serve as "controls" and receive only Montanide ISA51 mixed with saline. The vaccine is injected into the muscle of the upper arm. Subjects are monitored for 30 minutes after each injection for possible side effects and take home a diary card to record their temperature and any symptoms that may appear over the next 13 days.

A blood sample is drawn before and on several occasions after each vaccination to check the subject's health and to evaluate the immune response to the vaccine. At 1, 3, 7, 14, and 21 days after each vaccination, participants come to the clinic for a check of vital signs (temperature, pulse, respiration, and blood pressure), brief physical examination, and history of symptoms since the previous visit.

DETAILED DESCRIPTION:
The purpose of this Phase 1 clinical trial is to evaluate the safety, reactogenicity and immunogenicity of two malaria transmission-blocking vaccines, PpPfs25 and ScPvs25, in healthy adult volunteers. Of the four species of malaria that infect humans, Plasmodium falciparum is responsible for the majority of these deaths. However, outside of Africa, most of the malaria is caused by Plasmodium vivax; although these cases result in few deaths, they represent a major cause of morbidity and lead to a significant impact on the quality of life. The development of a safe and effective vaccine that prevents the transmission of P. falciparum or P. vivax would be an important addition to the current methods for controlling the spread of malaria parasites. A vaccine designed to prevent oocyst development in the mosquito by eliciting transmission-blocking antibodies in the vertebrate host would protect other individuals in the vicinity from becoming infected from the immunized person. Thus, despite no immediate role in personal protection, transmission-blocking vaccines are a potentially powerful component of a multifaceted public health approach to controlling or eliminating malaria. This study will be conducted at the Johns Hopkins University - Bloomberg School of Public Health, Center for Immunization Research. Seventy-two healthy male and non-pregnant female volunteers ages 18-50 will be enrolled. This study will be single blinded (to volunteers) and placebo-controlled. The study will evaluate three dose levels of both the PpPfs25 and ScPvs25 malaria vaccines (5 microg, 20 microg, 80 microg) emulsified with Montanide ISA51 as compared to Montanide ISA51 given alone. Seventy-two volunteers (60 vaccine and 12 placebo) will be enrolled and assigned to one of six cohorts. In each cohort, 10 volunteers will receive vaccine and 2 will receive placebo. Volunteers will be vaccinated by intramuscular injection on days 0 and 120. The groups will be staggered such that adequate safety evaluation can be performed prior to dose escalation. The duration of the study is 18 months per volunteer. The primary objectives of this trial are to assess and compare, in a dose-escalating study, the safety and reactogenicity of the PpPfs25 and ScPvs25 transmission blocking vaccines as compared to adjuvant alone; and to assess and compare, in dose-escalating study, the duration of the antibody response over an 18 month period in each volunteer as well as the effect of boosting with a second vaccination at 4 months.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males or females between 18 and 50 years, inclusive.
* Good general health as a result of review of medical history and/or clinical tests at screening.
* Available for the duration of the trial (78 weeks).
* Willingness to participate in the study as evidenced by signing the informed consent document.

EXCLUSION CRITERIA:

* Pregnancy as determined by a positive urine human chronic gonadotrophin (B-hCG), if female.
* Volunteer unwilling to use reliable contraception methods for the duration of the trial, if female. (Reliable methods of birth control include: pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, abstinence, and post-menopause)
* Currently breast-feeding (if female).
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.
* Laboratory evidence of liver disease (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] greater than the upper limit of normal of the testing laboratory).
* Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory).
* Laboratory evidence of hematologic disease (absolute neutrophil count less than 1,500/mm(3); hemoglobin less than the lower limit of normal of the testing laboratory, by sex; or platelet count less than 140,000/mm(3)).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis (greater than trace protein, or any glucose on urine dip will be confirmed negative prior to enrollment).
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Positive ELISA and confirmatory Western blot tests for HIV-1.
* Positive ELISA and confirmatory immunoblot tests for HCV.
* Positive HBsAg by ELISA.
* Known immunodeficiency syndrome.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study or while the study is ongoing.
* Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
* History of a surgical splenectomy.
* Receipt of blood products within the past 6 months.
* Previous receipt of an investigational malaria vaccine.
* History of a known allergy to nickel.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0
Dates: Start 2005-03-07; Study Completion 2008-06-17

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins School of Public Health, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Limsuwan A, Churdboonchart V, Moss RB, Sirawaraporn W, Sutthent R, Smutharaks B, Glidden D, Trauger R, Theofan G, Carlo D. Safety and immunogenicity of REMUNE in HIV-infected Thai subjects. Vaccine. 1998 Jan-Feb;16(2-3):142-9. doi: 10.1016/s0264-410x(97)88327-2. PMID 9607022
- [Derived] Wu Y, Ellis RD, Shaffer D, Fontes E, Malkin EM, Mahanty S, Fay MP, Narum D, Rausch K, Miles AP, Aebig J, Orcutt A, Muratova O, Song G, Lambert L, Zhu D, Miura K, Long C, Saul A, Miller LH, Durbin AP. Phase 1 trial of malaria transmission blocking vaccine candidates Pfs25 and Pvs25 formulated with montanide ISA 51. PLoS One. 2008 Jul 9;3(7):e2636. doi: 10.1371/journal.pone.0002636. PMID 18612426